CLINICAL TRIAL: NCT01046071
Title: The Analgesic Efficacy of Transversus Abdominis Plane Block After Laparoscopic Cholecystectomy: A Randomized Controlled Trial
Brief Title: The Analgesic Efficacy of Transversus Abdominis Plane Block After Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Pernille Lykke Petersen, MD, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM1-plp-09; 2009-017420-75 (EudraCT Number)
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2011-11-18 (Estimated); Status verified 2011-11

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: Transversus abdominis plane block, postoperative pain.
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- transversus abdominis plane block (Experimental): transversus abdominis plane block with ropivacaine
  Interventions: Procedure: transversus abdominis plane block
- block with saline (Placebo Comparator): 20 ml of isotonic saline bilateral
  Interventions: Procedure: TAP block placebo

INTERVENTIONS:
Procedure: transversus abdominis plane block — UL-guided TAP block with 20 ml of ropivacaine 0,5% bilateral, single dose.
  Other Names: Naropine; Postoperative pain; UL-guided nerve block
  Arms: transversus abdominis plane block
Procedure: TAP block placebo — UL-guided TAP block with 20 ml of saline bilaterally, single dose.
  Other Names: placebo block
  Arms: block with saline

SUMMARY:
The purpose of this study is to determine whether Transversus abdominis plane block as part of a multimodal postoperative regimen is superior to control in analgesic efficacy after laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic cholecystectomy
* ASA 1-3
* BMI 18-35
* Written consent

Exclusion Criteria:

* Do not understand danish
* Drug allergy
* Pregnancy
* Alcohol or drug abuse
* Chronic pain with consumption of opioids
* Consumption of NSAID, COX2inhibitors or paracetamol within 24 hours before the investigation
* Infection at the needle site.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-03; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Pain during cough. | 0,2,4,6,8,24 hours postoperative
  Area under the curve (AUC)-pain during cough based on measurements at 0,2,4,6,8,24 hours postoperative.

SECONDARY OUTCOMES:
Pain during rest | 0,2,4,6,8,24 hours postoperative
  Area under the curve (AUC)-pain during rest based on measurements at 0,2,4,6,8,24 hours postoperative.
Total opioid consumption | 0-24 hours postoperative
  Morphine consumption 0-2 hours postoperative. Ketobemidone consumption 2-24 hours postoperative.
Postoperative nausea and vomiting | 0,2,4,6,8,24 hours postoperative
  Nausea scores (0-3) at 0,2,4,6,8,24 hours postoperative. The number of vomits 0-2, 2-4, 4-6, 6-8 and 8-24 hours postoperative
Sedation | 0,2,4,6,8,24 hours postoperative
  Sedation scores (0-3) at 0,2,4,6,8,24 hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Pernille L Petersen, MD, Principal Investigator — Glostrup University Hospital, Copenhagen
Locations (1):
- Glostrup University Hospital, Department of anesthesia, Glostrup Municipality, Denmark